CLINICAL TRIAL: NCT07403864
Title: Effects of Acute Partial Sleep Deprivation on Metabolic Health and Cognitive Function
Brief Title: Effects of Acute Sleep Deprivation on Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202412HM033
Record Dates: First submitted 2026-01-23; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Glucose Intolerance; Energy Expenditure; Vascular Stiffness; Cognition
Keywords: Partial sleep deprivation; Sleep loss; Physical inactivity; Exercise habits
MeSH Terms: conditions — Glucose Intolerance; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (Experimental): Participants will have an 8-hour sleep opportunity in the lab from 23:00 to 07:00.
  Interventions: Behavioral: Normal sleep
- Partial sleep deprivation (Experimental): Participants will have a 3-hour sleep opportunity in the lab from 03:00 to 07:00.
  Interventions: Behavioral: Partial sleep deprivation

INTERVENTIONS:
Behavioral: Normal sleep — Participants will have an 8-hour sleep opportunity in the lab from 23:00 to 07:00.
  Arms: Normal sleep
Behavioral: Partial sleep deprivation — Participants will have a 3-hour sleep opportunity in the lab from 03:00 to 07:00.
  Arms: Partial sleep deprivation

SUMMARY:
This study will investigate whether various types of regular exercise can provide protective effects against metabolic abnormalities induced by sleep restriction. It will examine responses related to metabolic health, cognitive function, energy expenditure, subjective feelings, and human behaviors, including physical activity and energy intake.

DETAILED DESCRIPTION:
Sleep disturbances are common among the Taiwanese population due to work-related stress, shift work, and academic demands. Poor sleep can impair glucose and lipid metabolism, increasing the risk of cardiovascular disease and type 2 diabetes. This study will investigate whether regular exercise can mitigate these adverse effects. The findings aim to inform diverse exercise intervention strategies tailored to different populations to reduce health risks associated with insufficient sleep.

Participants will be healthy adults aged 20 to 45, categorized according to their habitual activity levels.

1. Sedentary: fewer than 7,000 steps per day and no regular exercise in the past 6 months.
2. Regular Aerobic Exercise: Running or cycling at least 2-3 times per week for the past 6 months.
3. Regular Resistance Exercise: Resistance training performed at least 2-3 times per week for the past 6 months, with minimal aerobic training.

Eligible participants must have regular sleep habits (Pittsburgh Sleep Quality Index [PSQI] ≤ 5), stable body weight (±3% over the past 3 months), no chronic diseases, no smoking or drinking habits, and no special diets.

Prior to the first main trial, participants will complete assessments of V̇O2max and maximal muscle strength within 7 to 14 days before the main trials. They will also record one week of daily physical activity, sleep patterns (including bedtime and wake-up times), and diet (covering two weekdays and one weekend day) to ensure they meet the inclusion criteria.

Day 1:

Physical activity will be restricted to a minimum, with no exercise permitted. Participants may eat freely before 15:00; however, all food intake will be recorded to enable replication prior to the second main trial. Napping is not allowed. Participants will arrive at the laboratory between 18:30 and 19:00. Upon arrival, after a 20-minute rest period, baseline measurements will be conducted, including body composition, waist and hip circumference, vascular function, subjective questionnaires, heart rate variability, food preference, a 20-minute energy metabolism assessment, and cognitive function testing. Subsequently, a standardized dinner will be provided by the researchers and consumed within 25 minutes. Participants will be allowed to wash and prepare between 20:00 and 20:30. From arrival onward, participants will remain seated on the experimental bed throughout the entire laboratory session. Continuous Glucose Monitoring (CGM) will be installed on day 1. Participants will have either an 8-hour sleep opportunity in the laboratory from 23:00 to 07:00 (i.e., normal sleep trial) or a 3-hour sleep opportunity from 03:00 to 07:00 (i.e., partial sleep deprivation trial).

Day 2:

Participants will wake at 07:00. After completing personal hygiene, they will rest for 20 minutes to ensure full wakefulness. At 07:30, a 20-minute resting metabolic rate assessment will be conducted, alongside the collection of heart rate variability and muscle oxygen saturation data. Subsequently, pulse wave velocity measurement, cognitive function tests, and subjective questionnaires will be administered.

This will be followed by a 3-hour oral glucose tolerance test (OGTT), during which 75 g of glucose will be ingested, and muscle oxygen saturation will be continuously monitored. Capillary blood samples will be collected via finger prick at 0, 30, 60, 90, 120, 150, and 180 minutes, alongside continuous glucose monitoring. Resting gas exchange, heart rate variability, and pulse wave velocity will be measured every 60 minutes. Blood pressure and visual analogue scale assessments-including sleep, appetite, and mood-will be recorded every 30 minutes. Cognitive function will be evaluated every 90 minutes.

Upon leaving the laboratory, participants will receive a pedometer and wearable devices. They will be instructed to record their dietary intake (using a food scale and photographic records), sleep patterns, and glucose levels on the experimental day and for the subsequent four consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-45 years.
* Body Mass Index (BMI) between 18.5-27 kg/m².
* No sleep-related medical conditions and good sleep quality, defined as a Pittsburgh Sleep Quality Index (PSQI) score ≤ 5.
* Usual bedtime between 22:00-01:00, wake-up time between 06:00-09:00, with an average sleep duration of 7 to 9 hours; chronotype classified as "definitely not evening type" (score ≥ 42 on the Morningness-Eveningness Questionnaire), and no changes in sleep patterns over the past 3 months.
* Without any metabolic or cardiovascular diseases, and not using medications that could affect metabolic responses.
* No specific dietary habits, such as intermittent fasting or a ketogenic diet.
* Maintaining a stable weight (no self-reported weight change ± 3 kg) for at least 3 months.
* Resting blood pressure ≤ 130/80 mmHg.
* No smoking or excessive alcohol consumption.
* Not a shift worker.
* No international travel across time zones has occurred within the past 3 months.

Exclusion Criteria:

* Special diets (e.g., intermittent fasting, ketogenic diet)
* Recent injuries or contraindications to intense exercise.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | Baseline measurements and continuously at regular intervals throughout the 3-hour OGTT.
  Glucose responses during the 3-hour oral glucose tolerance test (OGTT)
Pulse wave velocity (PWV) | 0 (baseline), 60, 120 and 180 minutes during OGTT
  Pulse wave velocity assessments (i.e., meters per second) will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Cognitive function (Accuracy) | 0 (baseline), 90 and 180 minutes during OGTT
  Accuracy (i.e., %) in computerized tests will be tested before and during the 3-hour oral glucose tolerance test (OGTT).
Cognitive function (Reaction time) | 0 (baseline), 90 and 180 minutes during OGTT
  Reaction time (i.e., milliseconds) in computerized tests will be tested before and during the 3-hour oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Resting energy expenditure | 0 (baseline), 60, 120 and 180 minutes during OGTT
  Energy expenditure will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Carbohydrate oxidation | 0 (baseline), 60, 120 and 180 minutes during OGTT
  Carbohydrate oxidation will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Fat oxidation | 0 (baseline), 60, 120 and 180 minutes during OGTT
  Fat oxidation will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Heart rate variability | 0 (baseline), 60, 120 and 180 minutes during OGTT
  Heart rate variability will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Muscle oxygen saturation | 0 minute (baseline) and throughout the entire 3-hour OGTT
  Muscle oxygen saturation data will be collected before and during the 3-hour oral glucose tolerance test (OGTT).
Blood pressure | 0 (baseline), 30, 60, 90, 120,150 and 180 minutes during OGTT
  Blood pressure (mmHg) assessments will be collected before and during the 3-hour oral glucose tolerance test (OGTT).